CLINICAL TRIAL: NCT07073209
Title: PENG vs Femoral Block for Hip Fracture, A Pragmatic Cluster-Randomized Study
Brief Title: PENG vs Femoral Block for Hip Fracture Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-07027709
Record Dates: First submitted 2025-06-25; First posted 2025-07-18 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hip Fractures
Keywords: Pain; Anesthesia; Analgesia; Hip Fracture; Peripheral nerve block; Regional Anesthesia
MeSH Terms: conditions — Hip Fractures; Pain; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Single-center, cluster-randomized, crossover trial.
  The crossover is not at an individual level in regard to the subjects but instead will be for the institutional policy regarding the block administration. A randomized schedule will be created for the type of block administered each month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG Block Administration (Experimental): Policy for the administration of the PENG block as per clinical guidelines to all subjects presenting to the hospital with a diagnosis of hip fracture and consenting to analgesic block
  Interventions: Procedure: PENG Block Administration; Drug: Bupivacaine , epinephrine Dexamethasone
- Femoral Block Administration (Experimental): Policy for the administration of the Femoral block as per clinical guidelines to all subjects presenting to the hospital with a diagnosis of hip fracture and consenting to analgesic block
  Interventions: Procedure: Femoral Block Administration; Drug: Bupivacaine , epinephrine Dexamethasone

INTERVENTIONS:
Procedure: PENG Block Administration — Policy for the PENG block administration:
  30 mL of Bupivacaine 0.25% 1:200,000 epinephrine Dexamethasone 4 mg%
  While these drugs are administered to participants, the intervention under evaluation is the PENG Block anesthesia technique.
  Arms: PENG Block Administration
Procedure: Femoral Block Administration — Policy for the Femoral block administration:
  30 mL of Bupivacaine 0.25% 1:200,000 epinephrine Dexamethasone 4 mg
  While these drugs are administered to participants, the intervention under evaluation is the Femoral Block anesthesia technique.
  Arms: Femoral Block Administration
Drug: Bupivacaine , epinephrine Dexamethasone — 30 mL of Bupivacaine 0.25% 1:200,000 epinephrine Dexamethasone 4 mg%

SUMMARY:
This study aims to compare the Pericapsular Nerve Group (PENG) block with femoral block for hip fracture pain. Participants presenting to the hospital with a diagnosis of hip fracture and consenting to analgesic block will receive either a PENG or femoral block. The choice of block will be dictated by a randomized monthly schedule, and all participants presenting during each four-week period will receive the designated block. A sub-group analysis will be performed to determine any difference in efficacy in participants with intracapsular versus extracapsular fractures.

DETAILED DESCRIPTION:
Each year, 250,000 adults in the US and 1.6 million worldwide suffer hip fractures. Peripheral nerve blocks, including femoral blocks, administered soon after admission to patients presenting with hip fractures have been shown to produce clinically and statistically significant reductions in pain scores, opioid consumption, the incidence of confusional state, and the time to mobilization.

Historically, lower extremity blocks for hip fracture pain have targeted the femoral nerve. The PENG block is a relatively novel ultrasound guided block that was first described in 2018 as an alternative to the more traditional femoral block for regional hip analgesia in hip fracture patients. The PENG block targets articular branches of the obturator nerve and accessory obturator nerve, as well as branches of the femoral nerve, the combination of which richly innervate the anterior hip capsule. In a case series of 5 patients presenting to the Emergency Department with hip fracture pain, the PENG block was demonstrated to be an effective nerve block for hip analgesia by reducing the numerical rating scale pain scores by 7 points on a 10 point scale. A larger study compared the PENG block to placebo, also in hip fracture patients presenting to the Emergency Department, and demonstrated a significant decrease of 3 in the dynamic NRS pain score at 1 and 3 hours post-block. A Cochrane review in 2017 demonstrated femoral blocks to have a 3.4 point reduction in pain scores compared to placebo. No study to date has compared the PENG block to the femoral block for acute hip fracture pain.

This study aims to compare the PENG block with femoral block for acute hip fracture pain in patients upon presentation who have not undergone surgical repair. Patients presenting to the hospital with a diagnosis of hip fracture and consenting to analgesic block will receive either a PENG or femoral block. The choice of block will be dictated by a randomized monthly schedule, and all patients presenting during each four-week period will receive the designated block. The primary outcome will be the change in NRS pain score from pre-block to one-hour post-block. Secondary outcomes will include NRS pain scores and opioid consumption for 24 hours post-block. A sub-group analysis will be performed to determine any difference in efficacy in patients with intracapsular versus extracapsular fractures.

This will be a pragmatic study with a multiple crossover cluster-controlled design. In this type of trial an intervention is implemented for all patients for a limited period of time and then substituted with the alternate intervention for a comparable amount of time. The order of intervention will be randomized. The repetition of the study periods, especially if conducted over a period of a year of more, has the effect of reducing time-dependent confounding from background improvements in healthcare and regression to the mean. The Hawthorne effect will be limited in this particular case because both of the interventions are already routinely and interchangeably used in our current practice for hip fracture analgesia. Research consent is usually waived in this type of trial design because the treatment received by subjects is identical to standard care and the exposure within a subject population is based only on time period rather than patient characteristics or consent.

As per current standard of care, all hip fracture patients admitted Monday - Friday, 7AM - 5PM, will be offered an analgesic lower extremity peripheral nerve block. Each month of the study will be randomized to either PENG or femoral block. All patients who consent to a block during each month will receive the designated block.

Data will be collected from the electronic medical record (EMR).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. ASA Classification 1-4
3. Documentation of a hip fracture diagnosis along with radiologic read indicating fracture location
4. Written, informed consent for analgesic peripheral block placement

Exclusion Criteria:

1. Altered mental status to the extent that it limits ability to report pain score
2. Patient or health care proxy refusal of analgesic nerve block
3. Allergy to study medications or contraindication to peripheral nerve block
4. Chronic pain diagnosis on preoperative opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Numerical Rating Scale (NRS) Pain Score One Hour Post Block for all Subjects | Baseline, 1-hour post block
  The Numerical Rating Scale (NRS) measures the intensity of pain a subject experiences. where subjects rate their pain on a scale from zero to ten and each number corresponds to a different level of intensity. The lowest score 0 represents no pain and the highest score 10 represents the most intense feeling of pain.
Mean Change in Numerical Rating Scale (NRS) Pain Score One-Hour Post Block in Intracapsular Hip Fractures | Baseline, 1-hour post block
  The Numerical Rating Scale (NRS) measures the intensity of pain a subject experiences. where subjects rate their pain on a scale from zero to ten and each number corresponds to a different level of intensity. The lowest score 0 represents no pain and the highest score 10 represents the most intense feeling of pain.
Mean Change in Numerical Rating Scale (NRS) Pain Score One-Hour Post Block in Extracapsular Hip Fractures | Baseline, 1-hour post block
  The Numerical Rating Scale (NRS) measures the intensity of pain a subject experiences. where subjects rate their pain on a scale from zero to ten and each number corresponds to a different level of intensity. The lowest score 0 represents no pain and the highest score 10 represents the most intense feeling of pain.

SECONDARY OUTCOMES:
Mean NRS Pain Scores up to 24 Hours Post-block for all Subjects | 0-24 hours post block
  The Numerical Rating Scale (NRS) measures the intensity of pain a subject experiences. where subjects rate their pain on a scale from zero to ten and each number corresponds to a different level of intensity. The lowest score 0 represents no pain and the highest score 10 represents the most intense feeling of pain.
Mean NRS Pain Scores up to 24 Hours Post-block in Intracapsular Hip Fractures | 0-24 hours post block
  The Numerical Rating Scale (NRS) measures the intensity of pain a subject experiences. where subjects rate their pain on a scale from zero to ten and each number corresponds to a different level of intensity. The lowest score 0 represents no pain and the highest score 10 represents the most intense feeling of pain.
Mean NRS Pain Scores up to 24 Hours Post-block in Extracapsular Hip Fractures | 0-24 hours post block
  The Numerical Rating Scale (NRS) measures the intensity of pain a subject experiences. where subjects rate their pain on a scale from zero to ten and each number corresponds to a different level of intensity. The lowest score 0 represents no pain and the highest score 10 represents the most intense feeling of pain.
Number of Oral Morphine Equivalents Administered for all Subjects | 0-24 hours post block
  Milligrams of oral morphine equivalent opioid consumption up to 24 hours post-block.
  Non-morphine opioids will be converted to an equivalent morphine dosage in milligrams for comparison across both block types. Oral morphine equivalent dosages are calculated using: Wen RY et al. A Comparison of Institutional Opioid Equianalgesia Tools: A National Study. J Palliat Med. 2022;25:1686
Number of Oral Morphine Equivalents Administered in Intracapsular Hip Fractures | 0-24 hours post block
  Milligrams of oral morphine equivalent opioid consumption up to 24 hours post-block.
  Non-morphine opioids will be converted to an equivalent morphine dosage in milligrams for comparison across both block types. Oral morphine equivalent dosages are calculated using: Wen RY et al. A Comparison of Institutional Opioid Equianalgesia Tools: A National Study. J Palliat Med. 2022;25:1686
Number of Oral Morphine Equivalents Administered in Extracapsular Hip Fractures | 0-24 hours post block
  Milligrams of oral morphine equivalent opioid consumption up to 24 hours post-block.
  Non-morphine opioids will be converted to an equivalent morphine dosage in milligrams for comparison across both block types. Oral morphine equivalent dosages are calculated using: Wen RY et al. A Comparison of Institutional Opioid Equianalgesia Tools: A National Study. J Palliat Med. 2022;25:1686

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Tedore, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neuman MD, Feng R, Carson JL, Gaskins LJ, Dillane D, Sessler DI, Sieber F, Magaziner J, Marcantonio ER, Mehta S, Menio D, Ayad S, Stone T, Papp S, Schwenk ES, Elkassabany N, Marshall M, Jaffe JD, Luke C, Sharma B, Azim S, Hymes RA, Chin KJ, Sheppard R, Perlman B, Sappenfield J, Hauck E, Hoeft MA, Giska M, Ranganath Y, Tedore T, Choi S, Li J, Kwofie MK, Nader A, Sanders RD, Allen BFS, Vlassakov K, Kates S, Fleisher LA, Dattilo J, Tierney A, Stephens-Shields AJ, Ellenberg SS; REGAIN Investigators. Spinal Anesthesia or General Anesthesia for Hip Surgery in Older Adults. N Engl J Med. 2021 Nov 25;385(22):2025-2035. doi: 10.1056/NEJMoa2113514. Epub 2021 Oct 9. PMID 34623788
- [Background] Riddell M, Ospina M, Holroyd-Leduc JM. Use of Femoral Nerve Blocks to Manage Hip Fracture Pain among Older Adults in the Emergency Department: A Systematic Review. CJEM. 2016 Jul;18(4):245-52. doi: 10.1017/cem.2015.94. Epub 2015 Sep 10. PMID 26354332
- [Background] Ritcey B, Pageau P, Woo MY, Perry JJ. Regional Nerve Blocks For Hip and Femoral Neck Fractures in the Emergency Department: A Systematic Review. CJEM. 2016 Jan;18(1):37-47. doi: 10.1017/cem.2015.75. Epub 2015 Sep 2. PMID 26330019
- [Background] Scurrah A, Shiner CT, Stevens JA, Faux SG. Regional nerve blockade for early analgesic management of elderly patients with hip fracture - a narrative review. Anaesthesia. 2018 Jun;73(6):769-783. doi: 10.1111/anae.14178. Epub 2017 Dec 26. PMID 29278266
- [Background] Giron-Arango L, Peng P. Pericapsular nerve group (PENG) block: what have we learned in the last 5 years? Reg Anesth Pain Med. 2025 May 6;50(5):402-409. doi: 10.1136/rapm-2024-105427. PMID 38724271
- [Background] Guay J, Parker MJ, Griffiths R, Kopp S. Peripheral nerve blocks for hip fractures. Cochrane Database Syst Rev. 2017 May 11;5(5):CD001159. doi: 10.1002/14651858.CD001159.pub2. PMID 28494088
- [Background] Griffiths R, Babu S, Dixon P, Freeman N, Hurford D, Kelleher E, Moppett I, Ray D, Sahota O, Shields M, White S. Guideline for the management of hip fractures 2020: Guideline by the Association of Anaesthetists. Anaesthesia. 2021 Feb;76(2):225-237. doi: 10.1111/anae.15291. Epub 2020 Dec 2. PMID 33289066
- [Background] White SM, Altermatt F, Barry J, Ben-David B, Coburn M, Coluzzi F, Degoli M, Dillane D, Foss NB, Gelmanas A, Griffiths R, Karpetas G, Kim JH, Kluger M, Lau PW, Matot I, McBrien M, McManus S, Montoya-Pelaez LF, Moppett IK, Parker M, Porrill O, Sanders RD, Shelton C, Sieber F, Trikha A, Xuebing X. International Fragility Fracture Network Delphi consensus statement on the principles of anaesthesia for patients with hip fracture. Anaesthesia. 2018 Jul;73(7):863-874. doi: 10.1111/anae.14225. Epub 2018 Mar 6. No abstract available. PMID 29508382
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Lin X, Liu CW, Goh QY, Sim EY, Chan SKT, Lim ZW, Chan DXH. Pericapsular nerve group (PENG) block for early pain management of elderly patients with hip fracture: a single-center double-blind randomized controlled trial. Reg Anesth Pain Med. 2023 Nov;48(11):535-539. doi: 10.1136/rapm-2022-104117. Epub 2023 Apr 13. PMID 37055189
- [Background] Sessler DI, Myles PS. Novel Clinical Trial Designs to Improve the Efficiency of Research. Anesthesiology. 2020 Jan;132(1):69-81. doi: 10.1097/ALN.0000000000002989. PMID 31809323
- [Background] Ford I, Norrie J. Pragmatic Trials. N Engl J Med. 2016 Aug 4;375(5):454-63. doi: 10.1056/NEJMra1510059. No abstract available. PMID 27518663
- [Background] Wen RY, Atayee RS, Edmonds KP. A Comparison of Institutional Opioid Equianalgesia Tools: A National Study. J Palliat Med. 2022 Nov;25(11):1686-1691. doi: 10.1089/jpm.2021.0678. Epub 2022 May 13. PMID 35559657
- See also: PMID: 34623788 — https://pubmed.ncbi.nlm.nih.gov/34623788/
- See also: PMID: 26354332 — https://pubmed.ncbi.nlm.nih.gov/26354332/
- See also: PMID: 26330019 — https://pubmed.ncbi.nlm.nih.gov/26330019/
- See also: PMID: 29278266 — https://pubmed.ncbi.nlm.nih.gov/29278266/
- See also: PMID: 38724271 — https://pubmed.ncbi.nlm.nih.gov/38724271/
- See also: PMID: 28494088 — https://pubmed.ncbi.nlm.nih.gov/28494088/
- See also: PMID: 33289066 — https://pubmed.ncbi.nlm.nih.gov/33289066/
- See also: PMID: 29508382 — https://pubmed.ncbi.nlm.nih.gov/29508382/
- See also: PMID: 30063657 — https://pubmed.ncbi.nlm.nih.gov/30063657/
- See also: PMID: 37055189 — https://pubmed.ncbi.nlm.nih.gov/37055189/
- See also: PMID: 31809323 — https://pubmed.ncbi.nlm.nih.gov/31809323/
- See also: PMID: 27518663 — https://pubmed.ncbi.nlm.nih.gov/27518663/
- See also: PMID: 35559657 — http://pubmed.ncbi.nlm.nih.gov/35559657/